CLINICAL TRIAL: NCT00889642
Title: A Multicenter Double-Blind Randomized Placebo Controlled Two-Arm Study Evaluating the Safety and Efficacy of the Iontophoretic Administration of Lidocaine and Epinephrine Using Lidocaine Iontophoretic Drug Delivery System (IDDS) to Provide Local Anesthesia for Venipuncture in Healthy Adult Volunteer Subjects
Brief Title: Safety and Efficacy Study of an Iontophoretic Patch Containing Lidocaine and Epinephrine for Venipuncture in Healthy Adult Volunteers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dharma Therapeutics Inc. (Industry)
Responsible Party: Ron Berenson, Acting Medical Director, Dharma Therapeutics Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Dharma-NSCO3
Record Dates: First submitted 2009-04-27; First posted 2009-04-29 (Estimated); Last update posted 2009-06-23 (Estimated); Status verified 2009-06

CONDITIONS: Local Anesthesia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Active Comparator): Contains Lidocaine and Epinephrine
  Interventions: Device: Iontophoretic Drug Delivery System with Lidocaine/Epinephrine
- Placebo (Placebo Comparator): Contains Epinephrine
  Interventions: Device: Iontophoretic Drug Delivery System with Epinephrine

INTERVENTIONS:
Device: Iontophoretic Drug Delivery System with Lidocaine/Epinephrine — Active- 10.5% Lidocaine/0.179% Epinephrine
  Arms: Active
Device: Iontophoretic Drug Delivery System with Epinephrine — Placebo- 0.179% Epinephrine
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effectiveness of administering Lidocaine and Epinephrine using an iontophoretic device treatment to provide local anesthesia to healthy adult volunteer subjects undergoing venipuncture.

ELIGIBILITY:
Inclusion Criteria:

* Subjects may be of any race, either sex, and must be >18 years of age
* Healthy subjects as per medical screening
* Subjects must have intact, healthy skin (no tattoos, surgical scars, skin infections, etc.) where the iontophoresis treatment will be performed
* Subjects must be alert, oriented, mentally competent, and able to understand and comply with the requirements of the study
* Subjects must have signed and dated a written informed consent
* Female subjects of childbearing potential must have a negative pregnancy test result prior to the iontophoresis treatment

Exclusion Criteria:

* Subjects with a known allergy or sensitivity to lidocaine, epinephrine or other local anesthetics of the amide or ester type
* Subjects with a know sensitivity to any components (e.g. adhesives) of the IDDSSubjects who have undergone venipuncture in the treatment area within the prior 2 weeks or longer if bruising or hematoma is apparent
* Subjects who have taken an analgesic pain medication during the 24-hour period prior to the venipuncture in the posterior surface of the hand
* Subjects with skin allergies or have skin diseases (e.g. psoriasis, eczema
* Subjects with an open skin lesion at the treatment site
* Subjects who are pregnant or breastfeeding
* Subjects exposed to an investigational drug or device within the past 30 days or are involved concurrently in other treatment clinical trials
* Subjects who participated in previous DTI/Transcu clinical studies related to this product
* Subjects with known concurrent illness
* Subjects with "current" known/admitted substance abuse (alcohol/drug)
* Subjects with pacemakers and/or externally mounted electronic devices
* Current or history of conditions that contraindicate use of iontophoretic treatment or venipuncture

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2009-05; Primary Completion 2009-05 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Following the iontophoresis treatment an IV will be inserted into the treatment area and the amount of pain will be assessed using the median visual analog pain scale (VAS). | 4 hours
Monitor the nature and frequency of adverse events associated with the iontophoretic device through observation during treatment. | 4 hours

SECONDARY OUTCOMES:
Determining the duration of anesthesia through standard pin prick testing. | 4 hours

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Advanced Clinical Research Institute, Anaheim, California
  - Vince & Associates Clinical Research, Overland Park, Missouri